CLINICAL TRIAL: NCT05374005
Title: The Impact of Excessive Dietary Sodium on Brain Health: Examining a Common But Neglected Risk Factor
Brief Title: The Impact of Excessive Dietary Sodium on Brain Health
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Bonnie Yin Ka LAM, Research Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2022.147
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Small Vessel Disease
Keywords: CSVD
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sporadic cerebral small vessel disease (CSVD) is not only the most common subtype of vascular dementia, in recent multi-center study showed that sporadic CSVD harbors in a third of Alzheimer's disease (AD) patients in 9 Asian regions. The CSVD increases the severity of cognitive impairment in these patients and has an etiological contribution to the development of AD. Studies demonstrated that CSVD is more prevalent in Chinese than in Australians and this association was independent of traditional vascular risk factors (e.g. hypertension). Other factors such as lifestyle, environmental or genetic factors may explain this difference. Although hypertension is an important cause for CSVD, it only accounts for a small proportion of the variance in CSVD. Irrespective of the cause, it is currently believed that endothelial dysfunction of CSVD is the key pathophysiological mechanism of CSVD. Having an effective treatment of CSVD will have an enormous impact on the prevention of dementia.

Excessive dietary sodium is an established risk factor for cardiovascular diseases, including stroke. It is traditionally linked to its effects in raising blood pressure. The Department of Health advocated reducing salt intake for the prevention of hypertension, coronary heart disease, and stroke.

However, recent epidemiological studies suggest that it may have a direct effect on cardiovascular diseases independent of blood pressure. A recent animal study showed that excessive dietary sodium-induced cerebral endothelial dysfunction, resulting in cognitive impairment. Interestingly, endothelial dysfunction was related to an adaptive immune response in the gut. A clinical study conducted in the United Kingdom suggested excessive dietary sodium intake may promote CSVD

A clinical study conducted in the United Kingdom suggested excessive dietary sodium intake may promote CSVD by increasing WMH volume in the brain, independent of its effects on blood pressure. Notably, a few animal studies showed that the association between high dietary sodium and worse cognitive function in the absence of blood pressure changes. This pinpoints the important role of dietary sodium as an independent contributor to brain health and cognition.

This study aims to assess the association between dietary sodium, neuroimaging measures, and cognition in cerebral small vessel disease and controls during the 18-month follow-up.

DETAILED DESCRIPTION:
This study hypothesis that high dietary sodium is associated with CSVD-related neuroimaging measures such as reduced white matter hyperintensities, total brain volume, and white matter structural integrity. The second hypothesis is that high dietary sodium is associated with worse cognitive function. These associations may be more prominent in the CSVD group compared to the control group and is independent of blood pressure.

Subjects with severe CSVD (n =110) and healthy controls (n =110) will be recruited.

2 trials of 24 hour urine will be collected at baseline visit and 2 trials of 24 hour urine will be collected at 18 months.

Clinical assessment (e.g. mood, cognition, physical activities, gait etc.) will be assessed at baseline and 18 months.

2 trials of Brain MRI will be conducted at baseline and 18 month visit

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity,
* age between 55 and 80-year-old, and
* a primary language of Cantonese.
* Extra inclusion criteria for CSVD group:

  1. Age-Related White Matter Change (ARWMC) Scale of 2 or early 3 in FLAIR MRI;
  2. Modified Functional Ambulation Classification 5 or above;
  3. Montreal Cognitive Assessment (MoCA) score < 25;

Exclusion Criteria:

* Hypernatremia (Na >146mmol/L) or hyponatremia (Na <134 mmol/L) from screening blood test;
* With sodium supplement;
* Renal failure (stage 4 & 5) with glomerular filtration rate < 29;
* performed cardiac surgery or neurosurgery, with cardiac failure;
* Had major psychiatric diseases
* Contraindications for MRI.
* Dementia or MoCA score lower than 2nd percentile of the age and education adjusted cutoff ;
* Cerebral white matter changes unrelated to neurodegenerative, e.g. CADASIL, X-linked adrenoleukodystrophy, metabolic diseases, multiple sclerosis, etc.|
* Contraindication to proposed imaging, e.g. chronic kidney disease (KDNIGO) stage 4 or above, acute kidney injury, hypersensitivity to gadolinium-based contrast, non-MRI conditional implants or prosthesis
* Medical condition that would not allow the patient to adhere to the protocol or complete the study.;
* Patient with established neurodegenerative disorders (e.g. Parkinson's Disease, Alzheimer's Disease, etc.);
* Pregnancy.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject with cSVD will be recruited at stroke unit and neurology clinic at Prince of Wales Hospital. Healthy volunteers will recruited through other community cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Change of level of urinary sodium | Baseline and 18 month
  24 hours of urine will be collected to measure the level of sodium
  The higher the sodium level the worse the outcome
Change of Gait | Baseline and 18 month
  Gait velocity will be assessed using the 8-meter walking time. Time for walking 8-m will be measured by a stopwatch. The faster of two trials will be used in the analysis
  The faster of the walking time the better outcome.
Change of balance | Baseline and 18 month
  Single leg stance time will be measured by asking participants, with their hands on their hips, to balance as long as possible on one leg with an upper limit of 30 seconds. Two trials for each leg will be performed. The best time of the four trials will be used for analysis. The longer the time duration the better outcome.
Change of Hong Kong MOntreal Cognitive Assessment | Baseline and 18 month
  Hong Kong MOntreal Cognitive Assessment (HK-MoCA) is a cognitive assessmenttool. Score from 0 to 30 . The lower score reflect the worse the outcome.
Change of The Chinese Geriatric Depression Scale 30 | Baseline and 18 month
  The Chinese Geriatric Depression Scale is used to detect depressive mood. Score 0 to 30. The higher the score, the worse the outcome
Change of Pittsburgh sleep quality index | Baseline and 18 month
  Pittsburgh sleep quality index Chinese Version is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The questionnaire contains frequency questions related to sleep quality, each question scale from 0 to 3. The higher the score, the worse the outcome. There is no total score available for this assessment
Change of Hong Kong List Learning Test | Baseline and 18 month
  Hong Kong List Learning Test is memory test in Chinese designed for the assessment of the processes and organizational strategies involved in learning verbal information. The more negative the standard deviation the worse the outcome
Food frequency questionnaire | Baseline
  The food frequency questionnaire serves the purpose of understanding the type of food that subject frequently consume in the past 12 months.
  There is no total score for this assessment. There is no positive and negative outcome available
Food frequency questionnaire | 18 month
  The food frequency questionnaire serves the purpose of understanding the type of food that subject frequently consume in the past 12 months.
  There is no total score for this assessment. There is no positive and negative outcome available
24 hour food intake | Baseline
  The 24 hour food intake serves the purpose of understanding the food that subject consume on the day of urine collection
  There is no positive and negative outcome available
24 hour food intake | 18 Month
  The 24 hour food intake serves the purpose of understanding the food that subject consume on the day of urine collection
  There is no positive and negative outcome available
Change of creatinine in urine | Baseline and 18 month
  24 hours of urine will be collected to measure the level of creatinine
  The higher the creatinine level the worse the outcome
change of urinary potassium | Baseline and 18 month
  24 hours of urine will be collected to measure the level of potassium
  The higher the potassium level the worse the outcome
Change of International Physical Activity Questionnaire | Baseline and 18 month
  the International Physical Activity Questionnaire is a self report assessment to investigate the daily activities (frequency, duration, and level) of subject within the 7 days prior assessment
  There is no total score available for this questionnaire. The higher duration and frequency and level of daily activities the better outcome
Change of Brain Peak Width of Skeletonized Mean Diffusivity | Baseline and 18 month
  Peak Width of Skeletonized Mean Diffusivity is a robust, fully-automated and easy-to-implement marker for cerebral small vessel disease based on diffusion tensor imaging, white matter tract skeletonization and histogram analysis. It is a biomarker for brain MRI images.

SECONDARY OUTCOMES:
Change of 24 hour blood pressure monitoring | Baseline and 18 Month
  Systolic and diastolic blood pressure will be measured using the 24-hour ambulatory blood pressure monitor. blood pressure will be measured at the same 24-hour period as urine measurement as blood

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Yin Ka Lam, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, N.T., Hong Kong

IPD SHARING:
Plan to Share IPD: No